CLINICAL TRIAL: NCT02167438
Title: Reducing Cesarean Childbirth Rates Using the Hem-Avert Perianal Stabilizer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Stetrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PB_004
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cesarean Section
Keywords: Cesarean; Section; second; stage; labor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational (Experimental): Application of the Hem-Avert device.
  Interventions: Device: Hem-Avert Perianal Stabilizer
- Control (No Intervention): No Application of the Hem-Avert device.

INTERVENTIONS:
Device: Hem-Avert Perianal Stabilizer
  Arms: Investigational

SUMMARY:
This study is being conducted to evaluate an FDA approved device called the HEM-AVERT® Perianal Stabilizer and the efficacy in reducing the C-section rate and/or reducing the second stage of labor times.

DETAILED DESCRIPTION:
Women may sometimes be reluctant to push resulting in a prolonged second stage labor, which could lead to a Cesarean section. This study will record the frequency of Cesarean sections in two groups to determine if there are any measurable differences.

The investigational device in this study is the HEM-AVERT® Perianal Stabilizer manufactured by Stetrix, Inc. This device has received previous FDA clearance as a Class II device to prevent hemorrhoids during childbirth. This study is being conducted by Stetrix, Inc. and falls within the guidelines set forth by the Food and Drug Administration in 21 CFR Section 812.2 as a non-significant risk study. The HEM-AVERT® Perianal Stabilizer is a Class II device in accordance with FDA regulation 21 CFR 890.5765. The Class II version of the device and the investigational device are identical in terms of materials, design, intended population and area used. The sole difference is that data will be collected in order to support an application to the FDA to obtain clearance of the device for the specific claim of reducing the C-section rate and/or reducing the second stage of labor times. This difference in data collection may be viewed as off-label use of the device although there is no new risk to the subject in the use of this device as an investigational device.

The primary objective of this study is to reduce the C-section rate and/or the second stage of labor times while using this device. For patients scheduled for a vaginal delivery, success is defined as completing the vaginal delivery process.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between the ages of 18 and 40 years old at the time of enrollment
2. Gestational age between 34 and 42 weeks at the time of enrollment
3. Live singleton gestation
4. Candidate for vaginal delivery.
5. Willing and able to comply with the study plan as indicated by understanding and signing the subject informed consent form

Exclusion Criteria:

1. Subject unable to speak English
2. Subject unable to understand and sign the informed consent form
3. Delivery planned outside the clinical center
4. Subject is scheduled for vaginal delivery with anticipated complications (i.e. including but not limited to non-vertex presentation or macrosomia >4,000 grams)
5. Subject scheduled for an elective cesarean birth
6. Preeclampsia with severe features, eclampsia, HELLP syndrome
7. Multiple Gestation
8. PROM (premature rupture of membranes)
9. Previous Cesarean Section
10. PTL (preterm labor)
11. Known major fetal anomaly or fetal demise.
12. Suspected or proven chorioamnionitis
13. Placenta previa
14. Maternal insulin dependent diabetes
15. Maternal health conditions deemed as risk factors by investigators such as renal or cardiopulmonary disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measuring the reduction in Cesarean section rates. | 12 Months
  This study is a single-site, prospective, randomized, concurrently-controlled study. Subjects will undergo screening to determine their enrollment eligibility. All subjects who meet inclusion criteria will be offered participation in this study.

SECONDARY OUTCOMES:
Measuring the reduction of second-stage of labor times. | 12 Months
  This is a single-site, prospective, randomized concurrently controlled study. Subjects will undergo screening to determine their enrollment eligibility. All subjects who meet inclusion criteria will be offered participation in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Francis Hospital, Memphis, Tennessee, United States